CLINICAL TRIAL: NCT01970826
Title: Sterilized Aseptic Versus Sterilized Clean Field for Dental Implant Placement - Randomized Clinical Control Trial for Non-inferiority Comparison
Brief Title: Compare Sterilized Clean vs Sterilized Aseptic Dental Implant Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Implantology Institute (Other)
Responsible Party: Principal Investigator, Andre Chen, Msc, Implantology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: II-05
Record Dates: First submitted 2013-10-19; First posted 2013-10-28 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Endosseous Dental Implant Failure; Bone Loss
Keywords: aseptic sterilized field; clean sterilized field; dental implants; Surgery
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Dental Implants; Time

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sterilized Clean Full-Mouth (Experimental): The operatory room will be prepared with clean instruments but with no aseptic preparation.
  Full-mouth dental implants placement will be made, Clean technique involves meticulous hand-washing, maintaining a clean environment by preparing a clean field, using clean gloves and sterile instruments, and preventing direct contamination of materials and supplies.
  There is contact between : non-sterile material in any change procedures and contact between sterile instruments or materials and any non-sterile surface or product.
  It will be evaluated the duration of surgery.
  Interventions: Procedure: Sterilized Clean; Procedure: Full-Mouth Dental Implants; Procedure: Duration of Surgery
- Sterilized Aseptic Full-Mouth (Active Comparator): The operatory room will be prepared with sterilized aseptic clean instruments. Full-mouth dental implants placement will be performed and involves meticulous hand washing, use of a sterile field, use of sterile gloves for application of a sterile dressing, and use of sterile instruments and fluid only. Involves the use of only sterile instruments and materials in dressing.
  There is no contact between : non-sterile material in any change procedures and contact between sterile instruments or materials and any non-sterile surface or products.
  It will be evaluated the duration of surgery.
  Interventions: Procedure: Sterilized Aseptic; Procedure: Full-Mouth Dental Implants; Procedure: Duration of Surgery
- Sterilized Clean Single (Experimental): The operatory room will be prepared with clean instruments but with no aseptic preparation.
  Single dental implants placement will be made, Clean technique involves meticulous hand-washing, maintaining a clean environment by preparing a clean field, using clean gloves and sterile instruments, and preventing direct contamination of materials and supplies.
  There is contact between : non-sterile material in any change procedures and contact between sterile instruments or materials and any non-sterile surface or products.
  It will be evaluated the duration of surgery.
  Interventions: Procedure: Single Dental Implants; Procedure: Sterilized Clean; Procedure: Duration of Surgery
- Sterilized Aseptic Single (Active Comparator): The operatory room will be prepared with clean instruments but with no aseptic preparation.
  Single dental implants placement will be made, Clean technique involves meticulous hand-washing, maintaining a clean environment by preparing a clean field, using clean gloves and sterile instruments, and preventing direct contamination of materials and supplies.
  There is contact between : non-sterile material in any change procedures and contact between sterile instruments or materials and any non-sterile surface or product.
  It will be evaluated the duration of surgery.
  Interventions: Procedure: Single Dental Implants; Procedure: Sterilized Aseptic; Procedure: Duration of Surgery
- Sterilized Clean - Partial (Experimental): The operatory room will be prepared with clean instruments but with no aseptic preparation.
  One or more dental implants will be made for partial rehabilitation, Clean technique involves meticulous hand-washing, maintaining a clean environment by preparing a clean field, using clean gloves and sterile instruments, and preventing direct contamination of materials and supplies.
  There is contact between : non-sterile material in any change procedures and contact between sterile instruments or materials and any non-sterile surface or product.
  It will be evaluated the duration of surgery.
  Interventions: Procedure: Sterilized Clean; Procedure: Partial Rehabilitation; Procedure: Duration of Surgery
- Sterilized Aseptic - Partial (Active Comparator): The operatory room will be prepared with clean instruments but with no aseptic preparation.
  One or more dental implants will be made for partial rehabilitation, Clean technique involves meticulous hand-washing, maintaining a clean environment by preparing a clean field, using clean gloves and sterile instruments, and preventing direct contamination of materials and supplies.
  There is contact between : non-sterile material in any change procedures and contact between sterile instruments or materials and any non-sterile surface or product.
  It will be evaluated the duration of surgery.
  Interventions: Procedure: Sterilized Aseptic; Procedure: Partial Rehabilitation; Procedure: Duration of Surgery

INTERVENTIONS:
Procedure: Single Dental Implants — place single unit dental implants, 2 mm below crestal bone and follow manufacturer guidelines.
  Other Names: Dental Fixtures
  Arms: Sterilized Aseptic Single; Sterilized Clean Single
Procedure: Sterilized Aseptic — Operatory room will be prepared totally aseptic
  Other Names: aseptic operatory room
  Arms: Sterilized Aseptic - Partial; Sterilized Aseptic Full-Mouth; Sterilized Aseptic Single
Procedure: Sterilized Clean — Operatory room will be prepared clean but not aseptic
  Other Names: Clean operatory room
  Arms: Sterilized Clean - Partial; Sterilized Clean Full-Mouth; Sterilized Clean Single
Procedure: Full-Mouth Dental Implants — dental implants for full-mouth implant rehabilitation.
  Other Names: Full-mouth rehabilitation; Full mouth implant supported rehabilitation
  Arms: Sterilized Aseptic Full-Mouth; Sterilized Clean Full-Mouth
Procedure: Partial Rehabilitation — two or more implants to support partial rehabilitation
  Other Names: partial implant-supported rehabilitation
  Arms: Sterilized Aseptic - Partial; Sterilized Clean - Partial
Procedure: Duration of Surgery — it will be measure the amount of time to perform the dental implant surgery. It will be measured from the time that the surgeon does the first incision until the last suture is made.
  Other Names: Time for implant placement

SUMMARY:
In patients that require dental implants , does performing the surgery in clean sterile field compared to aseptic field, produces more post-operatory complications, implant morbidity or patient discomfort ?

DETAILED DESCRIPTION:
The investigators intend to compare two types of operatory room preparation (aseptic versus clean), used world wide, for placing dental implants.

The investigators want to see if it has impact on post-operatory healing, osseointegration and success rate of dental implants.

Before Study begins the investigators will perform inter-observer agreement in surgical preparation of the surgical suite, implant placements and operatory-room behavior.

ELIGIBILITY:
Inclusion Criteria:

* All surgeries schedule for implant placement

Exclusion Criteria:

* Surgeries not made with local anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Post-Operatory Complications | From Implant Placement (Baseline) to 4 weeks after (T1)
  Measure the amount of adverse effects in both groups (aseptic vs clean) that happen between time frame baseline to 4 weeks.
Osseointegration | At 8 weeks (T2) after Baseline
  Measure the ability of dental implants to integrate into bone in both groups (aseptic vs clean)

SECONDARY OUTCOMES:
Marginal bone loss | At Final Restoration placement - Expected Average of 12 Weeks after baseline
  measure the amount of marginal bone loss at the time of final restoration placement
Patient Satisfaction | At 2 weeks
  measure the amount of post-operatory discomfort of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Andre Chen, Msc, Principal Investigator — University of Lisbon, College of Dentistry; João Caramês, Phd, Study Director — University of Lisbon, College of Dentistry; João Canta, Msc, Study Chair — University of Lisbon, School of Dentistry; Helena Francisco, Msc, Study Chair — University of Lisbon, College of Dentistry
Locations (1):
- University of Lisbon, School of Dentistry, Lisbon, Lisbon District, Portugal